CLINICAL TRIAL: NCT03826355
Title: Impact on Ovarian Reserve According to the Type of Ovarian Endometrioma Excision: Laser Versus Conventional Cystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Francisco Carmona, Head of Gynecology, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OR
Record Dates: First submitted 2019-01-20; First posted 2019-02-01 (Actual); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Endometriosis Ovary
MeSH Terms: interventions — Carbon Dioxide

STUDY DESIGN:
Intervention Model Description: Randomized prospective pairwise-data study. Patients with bilateral endometrioma with surgical indication will be selected. Ovarian reserve will be evaluated before and after surgery in both ovaries separately, using antral follicle count (AFC) and volume measurement. Type of surgery in each ovary will be randomized in the operating room (standard cystectomy vs laser vaporisation). A blinded ultrasonographer will evaluate AFC and volume measurement in both ovaries, before and three and six months after surgery. Therefore, each ovary will be compared with its contralateral in the same patient.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The ultrasonographer will be blinded to the procedure performed in each ovary after surgery. The patient will not be told which procedure has been performed in each ovary. The investigator will not know which procedure has been performed in each ovary until the end of the study. Only the surgeon will know which procedure is performed in each ovary.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stripping technique (Active Comparator): The endometrioma is removed according to standard surgery.
  Interventions: Procedure: Stripping technique
- Laser technique (Experimental): The endometrioma is drained, everted and then the inner wall of the endometrioma is vaporised with CO2 laser
  Interventions: Procedure: CO2 (carbon dioxide) laser vaporisation

INTERVENTIONS:
Procedure: CO2 (carbon dioxide) laser vaporisation — CO2 (carbon dioxide) laser is used to vaporise the inner wall of the endometrioma
  Arms: Laser technique
Procedure: Stripping technique — Identification of a cleavage plane and perform the cystectomy removing all the wall of the endometrioma from the healthy ovarian tissue
  Arms: Stripping technique

SUMMARY:
Endometriosis is a disease characterized by the presence of endometrial tissue outside the uterus cavity, causing important chronic pain and sterility in those patients suffering from it. It affects from 10 to 20% of women at reproductive age. Different types of endometriosis, which can coexist in the same patient, exist: deep infiltrating endometriosis (implants infiltrate > 5 mm the peritoneum), superficial endometriosis and ovarian endometriosis (OMA). OMA sometimes require surgery, and it is known that healthy ovarian tissue is also injured during resection. Consequently, ovarian reserve decreases, worsening the reproductive prognosis of patients affected. The main objective of the present study is to compare laser versus conventional OMA excision according to ovarian reserve in a pairwise-data study.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 45.
* Bilateral endometriomas.
* Endometrioma size > 3 cm.
* Pain and/or infertility as indication to surgical treatment.

Exclusion Criteria:

* History of cancer.
* Suspected malignancy.
* Evidence of premature ovarian failure.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Ovarian reserve | 7 months
  Antral follicular count by ultrasound: number of antral follicles.
Ovarian volume | 7 months
  Ovarian volume will be assesses by ultrasound, units given with milliliters

SECONDARY OUTCOMES:
Pregnancy rate | 6 months after surgery
  Pregnancy rate will be recorded during the 6 months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Carmona, MD PhD, Principal Investigator — Hospital Clinic of Barcelona

IPD SHARING:
Plan to Share IPD: No